CLINICAL TRIAL: NCT03551782
Title: An Open-label, Multicenter, Phase 1b Study of JNJ-63723283, a PD-1 Inhibitor, Administered in Combination With Apalutamide in Subjects With Metastatic Castration-Resistant Prostate Cancer
Brief Title: A Study of Cetrelimab (JNJ-63723283), a Programmed Cell Death Receptor-1 (PD-1) Inhibitor, Administered in Combination With Apalutamide in Participants With Metastatic Castration-Resistant Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR108476; 2018-000182-37 (EudraCT Number); 56021927PCR2032 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2018-05-30; First posted 2018-06-11 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Castration-Resistant Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms, Castration-Resistant | interventions — apalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1 (Experimental): Biomarker-negative or biomarker-unknown participants with adenocarcinoma (and not treatment-emergent small-cell neuroendocrine prostate cancer [t-SCNC]) who progressed on abiraterone acetate plus prednisone/prednisolone (AA-P) will be enrolled in this cohort. Participants will receive cetrelimab 480 milligram (mg) plus apalutamide 240 mg daily starting Cycle 1 (each cycle of 28 days).
  Interventions: Drug: Cetrelimab 480 mg; Drug: Apalutamide 240 mg
- Cohort 2 (Experimental): Biomarker-negative or biomarker-unknown participants with adenocarcinoma (and not t-SCNC) who progressed on apalutamide, darolutamide, or enzalutamide will be enrolled in this cohort. Participants will receive cetrelimab 480 mg plus apalutamide 240 mg daily starting Cycle 1.
  Interventions: Drug: Cetrelimab 480 mg; Drug: Apalutamide 240 mg
- Cohort 3 (Experimental): Biomarker-positive participants who progressed on AA-P will be enrolled in this cohort. Participants will receive cetrelimab 480 mg plus apalutamide 240 mg daily starting Cycle 1 (each cycle of 28 days).
  Interventions: Drug: Cetrelimab 480 mg; Drug: Apalutamide 240 mg
- Cohort 4 (Experimental): Biomarker-positive participants who progressed on apalutamide, darolutamide, or enzalutamide will be enrolled in this cohort. Participants will receive cetrelimab 480 mg plus apalutamide 240 mg daily starting Cycle 1 (each cycle of 28 days).
  Interventions: Drug: Cetrelimab 480 mg; Drug: Apalutamide 240 mg
- Cohort 5 (Experimental): Biomarker-negative participants with t-SCNC who progressed on treatment with AA-P, apalutamide, darolutamide, or enzalutamide will be enrolled in this cohort. Participants will receive cetrelimab 480 mg plus apalutamide 240 mg daily starting Cycle 1 (each cycle of 28 days).
  Interventions: Drug: Cetrelimab 480 mg; Drug: Apalutamide 240 mg

INTERVENTIONS:
Drug: Cetrelimab 480 mg — Cetrelimab 480 mg will be administered intravenously (IV) on Cycle 1 Day 1, then every 4 weeks thereafter (Q4W).
  Other Names: JNJ-63723283
Drug: Apalutamide 240 mg — Apalutamide 240 mg (4*60 mg) tablets per day will be administered orally.
  Other Names: JNJ-56021927

SUMMARY:
The purpose of this study is to evaluate the safety of the combination of cetrelimab, with apalutamide and to define a population of participants with metastatic castration-resistant prostate cancer (mCRPC) who respond to treatment with the combination of cetrelimab and apalutamide.

DETAILED DESCRIPTION:
This study is of participants originally diagnosed with adenocarcinoma of the prostate who have now developed mCRPC and who have progressed on therapy with abiraterone acetate plus prednisone/prednisolone (AA-P), apalutamide, darolutamide, or enzalutamide. Participants with treatment-emergent small-cell neuroendocrine prostate cancer (t-SCNC) assessed by the screening biopsy may be considered for this study. Participants must have confirmed prostate-specific antigen (PSA) progression per Prostate Cancer Clinical Trials Working Group (PCWG3) criteria. The primary hypothesis is that treatment with cetrelimab and apalutamide is safe and leads to improvement in the 12-week PSA response rate. The study consists of an Optional Pre-screening Period, Screening period (28 days prior to Cycle 1 Day 1), Treatment Period, End-of-Treatment Visit (performed after the last dose of study drug is administered), and Follow-up Period (participants will have Follow-up assessment every 12 weeks after the End-of-Treatment Visit). The efficacy, safety, and pharmacokinetics of cetrelimab in combination with apalutamide will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed adenocarcinoma of the prostate. Treatment-emergent small-cell neuroendocrine prostate cancer (t-SCNC) on screening biopsy may be eligible for cohort 5
* Metastatic disease as documented by technetium-99m (99mTc) bone scan or metastatic lesions by computed tomography (CT) or magnetic resonance imaging (MRI) scans (visceral or lymph node disease). CT-portion of positron emission tomography (PET)/CT scan may be used for eligibility. If lymph node metastasis is the only evidence of metastatic disease, it must be greater than (>=) 1.0 centimeter (cm) in the short axis and above the level of the iliac bifurcation
* Progressed while on therapy with abiraterone acetate plus prednisone/prednisolone (AA-P), enzalutamide, darolutamide, or apalutamide for mCRPC. No washout is required and no additional therapy may have been administered between discontinuation of AR-targeted the agent and study treatment. Participants will be assigned to cohorts based on the results of the biomarker panel. Cohort 1: Biomarker-negative or biomarker-unknown participants with adenocarcinoma (and not t-SCNC) who progressed on abiraterone acetate plus prednisone/prednisolone (AA-P); Cohort 2: Biomarker-negative or biomarker-unknown participants with adenocarcinoma (and not t-SCNC) who progressed on apalutamide, darolutamide, or enzalutamide; Cohort 3: Biomarker-positive participants who progressed on AA-P; Cohort 4: Biomarker-positive participants who progressed on apalutamide, darolutamide, or enzalutamide; Cohort 5: Biomarker-negative participants with t-SCNC who progressed on treatment with AA-P, apalutamide, darolutamide, or enzalutamide
* Surgical or medical castration, with testosterone levels of less than (<)50 nanogram per deciliter (ng/dL). If the participant is being treated with gonadotropin-releasing hormone (GnRH) analogs (participant who has not undergone bilateral orchiectomy), this therapy must have been initiated at least 4 weeks prior to first dose of study drug and must be continued throughout the study
* Eastern Cooperative Oncology Group Performance Status (ECOG) prostate-specific (PS) grade of 0 or 1

Exclusion Criteria:

* Initial diagnosis of primary prostatic neuroendocrine or small cell carcinoma
* Brain metastases
* Prior treatment with an anti-programmed cell death receptor-1 (PD-1), anti-programmed cell death ligand 1 (PD-L1), or anti-cytotoxic T-lymphocyte antigen 4 (CTLA-4) antibody
* Prior chemotherapy, except for docetaxel for hormone-sensitive prostate cancer (HSPC)
* Prior therapy with poly adenosine diphosphate (ADP)-ribose polymerase (PARP) inhibitors

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-06-28 (Actual); Primary Completion 2021-11-11 (Actual); Study Completion 2021-11-11 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs) | Approximately 2 years
  An AE is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Number of Participants with AEs by Severity | Approximately 2 years
  Severity of AEs will be assessed using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE). Any AE not listed in the NCI CTCAE will be graded according to the investigator clinical judgment by using the standard grades as follows: Grade 1 Mild: Awareness of symptoms that are easily tolerated, causing minimal discomfort and not interfering with everyday activities; Grade 2 Moderate: Sufficient discomfort is present to cause interference with normal activity; Grade 3 Severe: Extreme distress, causing significant impairment of functioning or incapacitation. Prevents normal everyday activities; Grade 4: Life-threatening or disabling AE; Grade 5: Death related to the AE.
Percentage of Participants with Prostate-Specific Antigen (PSA) Response at Week 12 | Week 12
  Percentage of participants with baseline in PSA level response (greater than or equal to [>=]50 percent [%] decrease from baseline in PSA) will be reported at Week 12.

SECONDARY OUTCOMES:
Maximal PSA Decline | Approximately 2 years
  Maximal PSA decline is defined as maximal percent decrease in PSA at any time during treatment.
Percentage of Participants with Circulating Tumor Cell (CTC) Response | Approximately 2 years
  Percentage of participants with CTC response (either CTC less than [<]5 cells/7.5 milliliter [mL] with CTC >=5 at baseline or CTC = 0 cells/7.5 mL with CTC >=1 at baseline) will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (34):
- United States (11):
  - University of California San Francisco (UCSF) - Prostate Cancer Center, San Francisco, California
  - Regional Urology LLC, Shreveport, Louisiana
  - University of Michigan Health System, Ann Arbor, Michigan
  - Washington University, Bay Saint Louis, Mississippi
  - New York University Langone Medical Center, New York, New York
  - Icahn School of Medicine at Mount Sinai - The Derald H. Ruttenberg, New York, New York
  - Levine Cancer Institute, Carolinas HealthCare System, Charlotte, North Carolina
  - Centers for Advanced Urology, LLC; d/b/a MidLantic Urology, Bala-Cynwyd, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Texas, MD Anderson Cancer Center, Houston, Texas
  - Virginia Oncology Associates, Norfolk, Virginia
- Belgium (2):
  - Grand Hôpital de Charleroi, site Notre Dame, Charleroi
  - AZ Maria Middelares, Ghent
- Canada (3):
  - Cross Cancer Institute, Edmonton, Alberta
  - University of Toronto, Toronto, Ontario
  - Centre de Recherche du CHUM, Montreal, Quebec
- Istituto Europeo di Oncologia Servizio Radioterapia, Milan, Italy
- Netherlands (3):
  - NKI-AVL, Amsterdam, Amsterdam
  - UMC Radboud, Nijmegen
  - Sint Franciscus Gasthuis, Rotterdam
- Russia (5):
  - Moscow City Clinical Hospital # 62, Moscow
  - Hertzen Oncology Research Institute, Moscow
  - Clinical Oncology Dispensary, Omsk
  - Non-State Healthcare Institution 'Road Clinical Hospital of Russian Railways', Saint Petersburg
  - Russian Scientific Center of Radiology and Surgical Technologies, Saint Petersburg
- Spain (9):
  - Hosp. Univ. Vall D Hebron, Barcelona
  - Hosp. Gral. Univ. Gregorio Marañon, Madrid
  - Hosp. Univ. Ramon Y Cajal, Madrid
  - Hosp. Univ. Fund. Jimenez Diaz, Madrid
  - Hosp. Univ. Hm Sanchinarro, Madrid
  - Hosp. Virgen de La Victoria, Málaga
  - Hosp. Quiron Madrid Pozuelo, Pozuelo de Alarcón
  - Hosp. Univ. Marques de Valdecilla, Santander
  - Instituto Valenciano de Oncologia, Valencia